CLINICAL TRIAL: NCT05421143
Title: Co-design of a Seamless Person-centered Intervention to Optimize Medication Use Across Healthcare Levels
Acronym: CIRCLE
Status: Recruiting | Type: Observational
Sponsor: Malin Olsen Syversen (Other)
Collaborators: Oslo University College (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, Malin Olsen Syversen, PhD student, Oslo University College
Organization: Oslo University College (Other)
Other Study IDs: 2536702
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Multimorbidity
Keywords: Person-Centered Care; Ethnography; Medications; Multiple long-term conditions; Self-efficacy; Patient preferences
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Quantitative study with medication reconciliation: The data collection will continue consecutively until the goal of 150 patients is reached. If it is feasible, we will try to reach 200 patients. We think 150-200 patients will give good insight into different types of medication discrepancies, since studies have shown that up to 90% of patients have at least one medication discrepancy in primary care.
- Qualitative semi-structured interviews with patients and next of kin: A selection of patients from the quantitative study described above will be chosen purposively and step by step along the way to ensure the informational strength in the selection. When possible, we will include next of kin in the interviews together with the patient. We aim to include around 20-30 patients, without counting in next of kin. The part will be accomplished together with the quantitative part. Every new interview will be compared with previous interviews to identify similarities and differences. Characteristics it is important to ensure variability for; women and men, different ethnicities, education type, spread in age, number of medications and help from next of kin/homecare nurses or not. It is also important to ensure variability in number and type of medications and diagnoses.
- Qualitative semi-structured interviews with HCP: HCP will be recruited purposively along the quantitative study to ensure the informational strength in the selection. We aim to include around 15-20 HCP. The HCP recruited are involved in the patients medication regime or management, this to ensure that they have knowledge about patients with multiple long term conditions. Every new interview will be compared with previous interviews to identify similarities and differences. Characteristics it is important to ensure variability for; woman and men, physicians and homecare nurses, spread in age, years of working experience, different ethnicities and number of medications the patients they care for use.

SUMMARY:
Multiple long term conditions entails various needs for complex medication treatment, which is a huge clinical challenge considering medication interactions and disease-medication interactions. It might affect quality of life, increase medical costs and needs, and cause patients to live several years with disabilities and reduced functional level. Multiple long term conditions is an important public health problem, since it is increasingly more common as the population is getting older.

It is well documented that communication problems exist between sectors in the healthcare system and that it creates an area of risk. There are many transfers that could be associated with risk for errors, as when patients are discharged from the hospital and is being transferred to the next level of care. When patients are discharged from the hospital, there is a need for transfer of correct information regarding medications. Transition of care leads to risk for medication discrepancies for the patients. Medication discrepancies are common within primary care and studies show that up to 90% of patients have at least one medication discrepancy in their lists. Different interventions have been tested to reduce medication discrepancies, but the interventions do not eliminate the need for medication reconciliations.

Higher patient satisfaction have been associated with improved patient safety, clinical effectiveness, health outcomes, adherence and lower resource utilization. According to Norwegian legislation, patients or users have a right to participate in the implementation of healthcare services, e.g. the choice between available and justifiable forms of service, examination methods and treatment methods. Person-centered care (PCC) is a concept that shifts the focus away from the traditional biomedical model to personal choice by applying shared decision-making. PCC reduce symptom burden, enhance patient activation, reduce readmission rates and improve quality of life.

Obtaining knowledge about medication discrepancies and perceptions from patients, next of kin and healthcare personnel (HCP) after the patient's hospital discharge could contribute to a better success rate for future interventions and services. It is therefore of interest to investigate which factors that are of importance for a successful seamless person-centered intervention to optimize medication use across healthcare levels. To obtain knowledge about medication discrepancies and perceptions, the study will include both quantitative and qualitative methods, and be using a design thinking framework. The persons included will represent a wide selection with respect to, among other things, age, gender, socio-economic background, profession and diagnoses. The patients, next of kin and HCP will be included after written, informed consent.

The aim of the project is to obtain knowledge about how the investigators can strengthen patient's self-efficacy and improve the information flow when it comes to medications, in the transition between the healthcare levels. To do so, the investigators need to identify facilitators and barriers to achieve a seamless medication treatment based on the user's needs. The results will form a basis for a new, improved intervention, which follow patients during the hospital stay and further out in the primary healthcare. The aim of this project is divided into the following parts:

* Investigate the frequency and type of medication discrepancies between the medication list in the discharge summary and medication use after hospital stay, to identify risk factors for which and why medication discrepancies occur in patients with multiple long term conditions.
* Map the perceptions of patients with multiple long term conditions and next of kin regarding medication use, shared decision-making and their opinions about previously published interventions to improve medication use.
* Evaluate HCP's perceptions regarding elements in patients with multiple long term conditions care that works well, what HCP believe do not work, with particular emphasis on the treatment with medications and transfer of care. In addition, how this care could be improved especially with the new intervention in mind.
* Using design thinking framework to create prototypes for a new intervention

Overall hypothesis for the project: Knowledge about medication discrepancies and perceptions from patients, next of kin and HCP regarding barriers and facilitators for a seamless medication treatment can contribute to an improved efficacy and implementation of the new, improved intervention.

DETAILED DESCRIPTION:
Our research group has previously completed the OPERA- and PERLE-studies, which explore the effect of a pharmacist intervention at the hospital and medication communication at hospital discharge from the patient perspective including the discharge process, respectively. The results from the PERLE-study gives a wider understanding of the discharge process and how patients experience medication communication at discharge. The results showed that every patient experienced a unique discharge process and that communication between healthcare personnel and patients was not sufficiently fostering patient empowerment and self-efficacy. The OPERA-study found no significant effect of the in hospital intervention on time to readmission or death within 12 months, but found a statistically significantly increased overall survival. The intervention in the OPERA-study consisted of clinical pharmacist added to the multidisciplinary treatment team working systematically according to the "Integrated Medicines Management" (IMM). IMM was originally developed in Northern Ireland and refined in Sweden. It is of importance to note that the model was used as without adaption to the Norwegian context and taking into account the traditional role for clinical pharmacists in Norwegian hospitals. This is especially related to the discharge process in which pharmacist would not normally be included.

Even though the OPERA-study showed statistically significant increased overall survival, is it desirable with a new intervention that fits better to the Norwegian context. Furthermore, a study suggest that medication reconciliation, medication review and post-discharge interventions should be performed all together as an integrated part of a multi-faceted program for better outcomes, and not isolated. This leads to a demand for a new intervention that extend beyond the hospital stay to achieve a seamless person-centered intervention to optimize medication use across healthcare levels. In designing the new intervention, the investigators need to obtain more knowledge about how to inform intervention development, study design and planning with respect to the user's needs. This is important since it is shown that patients are effective and willing contributors by supporting their own medication safety at transfers in the healthcare system. When developing a complex intervention, it is important to identify facilitators and barriers, e.g. to ensure that HCP involved in its delivery find it suitable and not in conflict with their daily tasks.

This study will use a design thinking framework based on the Three I's developed by IDEO: Inspiration, Ideation and Implementation. Inspiration focuses on learning how to better understand people to create possibilities, ideation focuses on making sense of that the investigators have heard to identify opportunities for design and generate ideas, and implementation focuses on bringing the investigators solutions to life to maximize its impact. This framework is a field guide to human-centered design as a way to apply design techniques to social service and innovation sectors, such as healthcare. This study will focus on the two first I's, namely the inspiration and ideation phase, whereas the third I, the implementation phase, will be covered in future projects.

The inspiration phase will comprise the following methods:

* Literature search to identify previously published models which might be suitable
* A quantitative part that assesses the number and type of medication discrepancies after hospital discharge by medication reconciliation
* A qualitative part in the form of semi-structured interviews and field notes including patients, next of kin and HCP

The investigators will focus on learning how to better understand people, and will use some of the aspects from the methodology of ethnography (38). Ethnographic research focuses on the social aspect of the research object. Ethnography is a multidimensional research approach covering a range of qualitative methods, including interviews and observations. Gathering ethnographic data is often termed doing fieldwork, with the field referring to the specific sites or locations where the data collection takes places. Using an ethnographic approach to understand aspect of medication use after newly being discharged could provide new, important insights to the field, both in theory development and to inform applied research projects.

The ideation phase will comprise the following methods:

The investigators will create personas and scenarios using the baseline understanding gathered from the inspiration phase. The created personas and scenarios will be further explored through workshops for prototyping. The workshops will aim to include relevant stakeholders, e.g. end users, comprising patients, next of kin and healthcare professionals (e.g. nurses, doctors and pharmacists), researchers and designers, together to work collectively during the prototyping.

The ideation phase will lead into the implementation phase for further planning of the future intervention.

Inspiration phase:

Literature search Before the inclusion starts, the investigators will perform a literature search through relevant research in PubMed and Medline, using search terms such as "patient-centered care", "person-centered care", "decision-making", "health communication", "self-efficacy", "medication management", "medication instructions", "patient participation", "patient preference", "patient transfer", "personal health records", "patient's drug list" and "electronic patient record". This to identify previously published models for an intervention.

Recruitment of study participants:

Participants to the quantitative and qualitative parts will be recruited simultaneously. Patients admitted to the Internal medicines ward and Geriatric ward, Oslo University Hospital (OUS), Ullevål, and a selection of their HCP and (if applicable) next of kin, will be included. Employees at the wards will ask inpatients for permission for one of the data collectors to inform and ask about participation in the study. This will take place close to the patients discharge (1-3 days ahead). Participants will be enrolled at the hospital, after written, informed consent. Consent from patients and next of kin will be obtained for medication reconciliation and interviews by use of one consent form. Consent will be obtained from HCP after their patient's enrollment in the study.

The data collection will take place face to face in the patient's home, HCP offices or other suitable location (e.g. meeting room at the hospital), approximately 1-2 weeks after the patients hospital discharge. A pilot study will be carried out during the spring 2022. The inclusion of patients, next of kin and HCP to the main study will start in the autumn 2022 and continue until the different parts have reach their goal, and for the qualitative parts; also have enough information power. The goal is to include patients, next of kin and HCP in the period from August 2022-July 2024. To further enrich the data, some patients might be selected for additional follow up interviews, after additional 3-4 weeks.

Number of persons to be included:

Quantitative study with medication reconciliation: The data collection will continue consecutively until the goal of 150 patients is reached. If it is feasible, the investigators will try to reach 200 patients. The investigators think 150-200 patients will give good insight into different types of medication discrepancies, since studies have shown that up to 90% of patients have at least one medication discrepancy in primary care. The inclusion and medication reconciliation will be done by the PhD-student together with master students in pharmacy.

Qualitative semi-structured interviews with patients and next of kin: The data collection will continue until the study have enough information power. This means that a selection of patients from the quantitative study described above will be chosen purposively and step by step along the way to ensure the informational strength in the selection. When possible, the investigators will include next of kin in the interviews together with the patient. The investigators aim to include around 20-30 patients, without counting in next of kin. For the follow-up interviews, approximately 5-8 patients will be selected. The part will be accomplished together with the quantitative part. Every new interview will be compared with previous interviews to identify similarities and differences. Characteristics it is important to ensure variability for; women and men, different ethnicities, education type, spread in age, number of medications and help from next of kin/homecare nurses or not. It is also important to ensure variability in number and type of medications and diagnoses. The inclusion and interviews of patients will be done by the PhD-student and master students in pharmacy.

Qualitative semi-structured interviews with HCP: The data collection will continue until the study have enough information power. This means that HCP will be recruited purposively along the quantitative study to ensure the informational strength in the selection. The investigators aim to include around 15-20 HCP. The HCP recruited are involved in the patients medication regime or management, this to ensure that HCP have knowledge about patients with multiple long term conditions. Every new interview will be compared with previous interviews to identify similarities and differences. Characteristics it is important to ensure variability for; woman and men, physicians and homecare nurses, spread in age, years of working experience, different ethnicities and number of medications the patients the HCP care for use. The inclusion and interviews of HCP will be done by the PhD-student.

Training and piloting:

Medication reconciliation and interviews will be done by the PhD-student and master students in pharmacy after receiving adequate training of clinical work. Training in medication reconciliation will be performed in accordance with procedures from the Hospital Pharmacies Enterprise, South-Eastern Norway, by an experienced clinical pharmacist. The procedure is based on the IMM-model for clinical pharmacists.

Both the PhD-student and master students will receive training and supervision in interviewing methodology from a researcher in the project group with strong competence in qualitative methods. During the spring 2022, the PhD-student will complete a course in qualitative research methods at the University of Oslo (UiO). The master students will complete relevant research preparatory courses during spring 2022.

The study procedures and documents will be piloted to obtain input to their finalization, e.g. the interview guide, and the practicability of the data collection tools. Inclusion of patients to the pilot will continue until sufficient feedback has been obtained. The inclusion to the pilot will follow the study criteria, as described above. If only minimal or no changes to the documents are deemed necessary, persons included to the pilot might be included in the study population described above. The pilot for all parts will start at the same time, and be finished when all details are in order. The PhD-student will have assistance from the research group for detailed design of the study during the pilot, and assistance as needed during the study. Consent to participate in the pilot study will be obtained as described above.

Instruments Quantitative study with medication reconciliation: The medication reconciliation will describe medication discrepancies between the medication list in the discharge summary and the actual medication use after hospital discharge. The medication discrepancies will be explored in conversation with the patient or, if the patient agrees to this, next of kin or other relevant information sources such as the GP or home-care nurse, to figure out why medication discrepancies have occurred. This could for example be changes done by the GP after hospital discharge. The medication reconciliation form from Hospital Pharmacies Enterprise, South-Eastern Norway (attached) will be used to do this task in accordance to their procedure for performing this (attached). The data will be analyzed consecutively to ensure that all details is included. A digital tool has been developed for the data collection in this study (attached).

Qualitative semi-structured interviews with patients and, if present, next of kin: The interviews will focus on patients and next of kin perceptions regarding medication use, shared decision-making when it comes to medications and their opinions about previously published interventions. Open questions will primarily be used in the interviews adjusted to each individual patient to explore different patient perspectives. The interview guide will be divided into themes and contain some predefined overarching questions with examples of possible probing questions. Furthermore, field notes will be taken to describe the setting, issues observed with relevance to the administration of medications, persons present and time consumption for the interviews. The interviews with patients and next of kin will focus on the following:

* How patients experience being a medication user, what patients think work and what patients think do not work. If something could be done to make medication use a more pleasant (rather than coercive) experience
* How patients use and assesses the utility value of digital solutions
* Experienced factors of PCC during the hospital stay, at discharge and after discharge, with a view to medication treatment
* Their opinions about previously published interventions with examples The interviews will be audiotaped, when the patients and (if present) next of kin agrees to this. If the patient does not consent to recording, notes will be taken. The interviewers will transcribe consecutively to prevent memory-bias, and to ensure that all details and own reflections comes with. The interviewers will read each other's transcripts and meet regularly to ensure the quality of the interviews. Follow-up interviews will be informal in nature, with no specific pre-defined interview guide.

Qualitative semi-structured interviews with HCP:

The interviews will focus on HCP's perceptions regarding factors, barriers and facilitators in the care for patients with multiple long term conditions with importance for a new, improved intervention. Open questions will primarily be used in the interviews adjusted to each individual HCP to explore different perspectives. The interview guide will be divided into themes and contain some predefined overarching questions with examples of possible probing questions. Furthermore, field notes will be taken to describe the setting and time consumption for the interviews.

The interviews with HCP will focus on the following:

* Factors in patients with multiple long term conditions medication treatment important for the patient's self-efficacy as a user of medicines and for their quality of life, both in a negative and positive direction, e.g. experience with patient empowerment and PCC
* How the system could improve with focus on digital solutions
* Their opinions about previously published interventions with examples The interviews will be audiotaped, when the HCP agrees to this. If the HCP does not consent, notes will be taken. The PhD-student will transcribe consecutively to prevent memory-bias (42), and to ensure that all details and own reflections comes with. The PhD-student will get help from the research group to read the transcripts and meet regularly to brief and discuss to ensure the quality of the interviews.

The main study for all parts will start at the same time, but the qualitative studies could be finished earlier if the investigators reach the goal of patients or HCP earlier than the goal in the quantitative study.

Data and measurement variables:

Demographic data and measurement variables will be retrieved from electronic patient record or directly from the patients and next of kin. Following data will be registered as part of inclusion about patients:

* Age
* Gender
* District in Oslo
* Profession
* Country of origin (if not Norwegian)
* Reason for admission
* Date for admission at the ward
* Multidose before admission (yes/no)
* Acute or elective admission
* Education level
* Cognitive function (if separate form has been filled in at the wards)
* Frailty scale (if separate form has been filled in at the wards)
* Assistance with medication administration before admission (manage themselves, manage themselves with help from next of kin or manage themselves with help from homecare nurses)

The following data will be collected as part of inclusion or interview about next of kin:

* Age
* Gender
* What kind of assistance next of kin give
* Education level
* Profession
* Relation to the patient
* How long next of kin have assisted the patient

The following data will be collected as part of inclusion or interview about HCP:

* Profession
* Age
* Gender
* Country of origin (if not Norwegian)
* Education level
* Years of working experience
* Years of working experience with patients with multiple long term conditions For patients, next of kin or HCP who do not consent to participate in the study, gender, age, role (patient, next of kin, HCP) and reason for refusal will be registered.

The following data will be collected consecutively after inclusion or at discharge for the patients:

* Type of ward the patient are discharged from
* Patients discharge summary
* Date of discharge
* Discharged to which care-level
* Medication list in the discharge summary: number of medications, ATC-code (level 5), medication name, dosage, formulation, regular/on demand use
* Diagnoses according to International Classification of Diseases (ICD) -10: Number and type, as described in the patients discharge summary
* Multidose after discharge (yes/no)
* Assistance with medication administration after discharge (manage themselves, manage themselves with help from next of kin or manage themselves with help from homecare nurses).

The following data will be collected during medication reconciliation:

* Complete medication use after discharge: In this way, the investigators will be able to count how many patients who has medication discrepancies and how many medication discrepancies each individual patients have. Why (if any) medication discrepancies have occurred.
* If the patient have assistance with medication administration: How much/type of help the patient have
* Descriptive data: Date, description of the setting, issues observed with relevance to the administration of medications, persons present and time consumption and information sources used during medication reconciliation.

Field work journal, field notes and other documents:

As part of the data collection process a fieldwork journal will be written by the data collectors. Here a narrative of the research process will be written down and form a basis for reflecting on the process and as inspiration for the data analysis. In addition, field notes will be written e.g. include impressions from the interviews, different kinds of observations done during the interviews, notes from the interviews. Information will also be collected from relevant documents, e.g. procedures from hospital and primary healthcare services.

Analyses:

Quantitative study: Medication reconciliation. Medication discrepancies revealed during medication reconciliation will be classified quantitatively, i.e. the proportion of patients with medication discrepancies, number of medication discrepancies per patient and type of medication discrepancies. In addition, the medication discrepancies will be categorized according to reasons why medication discrepancies have occurred.

Qualitative interviews and fieldwork. During the whole data collection process, field notes and fieldwork journal will be written by the data collectors. The interviews will be audiotaped, and will then be transcribed word for word. The interviews together with the field notes and journal will be analyzed inductively with inspiration from "content analysis" and/or systematic text condensation. The interviewers cooperate in the analyses to ensure quality, which means that the context is understood. Here also the field notes will be important in assuring reflectiveness of the process. Furthermore, the analyzes will focus on creating personas and scenarios for the ideation phase according to the design-thinking framework.

Ideation phase:

Workshops will be held with between six to eight participants comprising patients, next of kin, HCP (e.g. nurses, doctors and pharmacists), researchers and designers. Each workshop group will be assigned a scenario/personas and asked to conduct early prototyping. The prototyping will focus on supporting self-efficacy and transfer of medication information in the scenario. The output from the workshops together with the results of the inspiration phase, will be used by the research group to create models for the intervention. The created models for the intervention will be sent out by e-mail to previous participants in the inspiration- and ideation phases who are willing to contribute, for review and feedback.

Ethics The hypothesis of the project is that knowledge about medication discrepancies and perceptions from patients, next of kin and HCP after discharge can contribute to a better success rate for the new and improved intervention (29). Before the participants are included in the study, the participants will receive written information about the project and can decide for themselves whether they want to participate or not. It has been taken into account that some patients might refuse to participate, as the patients might not want to be visited by the study pharmacists, or that some might withdraw their consent. It will be acceptable that patients consent only to participate in the part with medication reconciliation, this can help to achieve our goal for this part of the study. Participants will be offered a small gift at maximum value of 100 Norwegian kroner, which is considered to small to influence their willingness to participate.

Information transfer when changing treatment level is a well known area of risk, and there is a need for greater focus on and knowledge about risk factors for medication discrepancies and perceptions of both patients, next of kin and HCP. The aim of the project is to form a basis for an improved intervention, which follows patients with multiple long term conditions during the hospital stay and through transition to the primary healthcare. This will be done by investigating medication discrepancies and map perceptions of patients, next of kin and HCP which, in both a positive and negative sense, are important for achieving seamless and person centered medication treatment, after the patients are discharged from hospital. It is expected that the results could give increased understanding that could contribute to a more seamless and person centered medication treatment in the future intervention and further development and improvement of healthcare services for patients.

Pharmacy students or the PhD-student, who are not affiliated with the internal medicines or geriatric wards on a daily basis, will perform the medication reconciliation, interviews and writing field notes. The pharmacy students and PhD-student are not involved in or have an overview of the overall picture and assessments behind decisions made regarding medication treatment. The pharmacy students and PhD-student have no active role in the treatment team and participation in the study thus does not contribute to any risk or harm for the participants beyond the time the participants spend on the medication reconciliation, interviews and/or workshop. No invasive procedures will be performed. If the medication reconciliation or interviews of the patients reveal critical discrepancies in the medication management in the patient's home, this will be passed on to the homecare nurse or GP.

Privacy and information:

The patients will be included after written, informed consent, see attachments. The same applies for HCP and next of kin. The attending physician determines whether the patients are competent to consent in those cases where there is doubt about this. After consent is obtained, the patient, next of kin or HCP will be given a study number. The included participants can at any time withdraw their consent, without having to give any justification for this. Registered data will be deleted if consent is withdrawn, as long as the data not yet has been included in the analysis work. Participants will receive a copy of the consent form. The signed consent forms will be kept in a locked filing cabinet in the project manager's office at UiO, and separate from the collected study data. The code list that connects patient identity to study number will be stored separately and secured from other data. The code list will be deleted no later than 10.01.2027.

All collected data will be treated confidentially and stored on the research server of UiO, Services for sensitive data (TSD). Data from medication reconciliation will be collected using a self-developed web form and stored directly on TSD. The interviews will be recorded on a Dictaphone and the audio files will be uploaded to TSD, immediately after the interview has ended. The interviews will be transcribed on TSD. The audio file will be deleted after the interview has been analyzed. Deidentified electronic research data will be processed using Statistical Package for the Social Sciences (SPSS) (quantitative data) or using Nvivo (qualitative data), on TSD.

The research project is approved by the Regional Committee for Medical and Health Research Ethics (420920/REK south-eastern C). In accordance with procedures for research at UiO, notification is sent and approved by the Norwegian Center for Research Data (NSD) (Ref. 919319).

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Adult ≥ 18 years
* Gives written, informed consent to participate in the study. If the patient is not competent to consent, consent can be obtained from the patient's next of kin.
* Residential address in Oslo
* Lives at home and normally manage their medications themselves (might have help from home-care nurses or next of kin)
* Scheduled to be discharged from the wards to their home or to short-term stay in nursing homes
* Uses at least four regular medications from at least two therapy classes (Anatomical Therapeutic Chemical (ATC) at first level

Health care personnel (HCP) and next of kin:

* Expected to be involved in the included patient's medication regime or management after hospital discharge
* Able and willing to give written, informed consent to participate in the study
* HCP should be general practitioners (GPs) or home-care nurses.

Exclusion Criteria:

Patients:

* Terminal and/or isolated due to infections
* Has previously been included in the study
* Has advanced cognitive failure, in accordance with assessment from treating physician
* Will not be discharged from the included wards to their homes (for example planned transfer to another ward or long-term stay at nursing home)
* Unable to communicate in Norwegian or English

HCP and next of kin:

* Unable to communicate in Norwegian or English
* HCP or next of kin that has previously been included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with multiple long-term conditions, their next of kin and HCP
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Frequency and type of medication discrepancies between the medication list in the discharge summary and medication use after hospital stay. | 2 years
  To identify risk factors for which and why medication discrepancies occur in patients with multiple long term conditions.

SECONDARY OUTCOMES:
Perceptions of patients with multiple long term conditions and next of kin | 1 year
  Regarding medication use, shared decision-making and their opinions about previously published interventions to improve medication use.
HCP's perceptions regarding elements in patients with multiple long term conditions care | 1 year
  What works well, what they believe do not work, with particular emphasis on the treatment with medications and transfer of care. In addition, how this care could be improved especially with the new intervention in mind.

CONTACTS AND LOCATIONS:
Overall Officials: Liv O Mathiesen, PhD, Study Director — University of Oslo; Malin O Syversen, Msc, Principal Investigator — University of Oslo
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Sharing in articles and after publishing. Anonymous data and transcripts.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publishing and before the data is deleted.
Access Criteria: For future research.